CLINICAL TRIAL: NCT04200560
Title: Autophagy Maintains Vascular Function Through a Novel Glycolysis-linked Pathway Regulating eNOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, John David Symons, Professor, University of Utah
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 00077971
Record Dates: First submitted 2019-06-18; First posted 2019-12-16 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Vascular Diseases
Keywords: Aging; Endothelial Cell Autophagy
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Adult Subjects (Experimental): Healthy adult subjects (18 - 30 years) will be assessed for markers of EC autophagy, eNOS activation, and NO generation before and after Rhythmic Handgrip Exercise
  Interventions: Other: Rhythmic Handgrip Exercise
- Healthy Older Adult Subjects (Experimental): Healthy older adult subjects (> 60 years) will be assessed for markers of EC autophagy, eNOS activation, and NO generation before and after Rhythmic Handgrip Exercise and after Chronic Exercise Training.
  Interventions: Other: Rhythmic Handgrip Exercise; Other: Chronic Exercise Training

INTERVENTIONS:
Other: Rhythmic Handgrip Exercise — 60 minute rhythmic handgrip exercise
Other: Chronic Exercise Training — Handgrip exercise training consisting of three 60-minute training sessions per week for eight weeks.
  Arms: Healthy Older Adult Subjects

SUMMARY:
Aging is inevitable and is the primary risk factor for developing cardiovascular disease. The molecular mechanisms that drive vascular dysfunction in the context of aging are incompletely understood. The overall hypothesis is that the age-related decline in endothelial cell (EC) autophagy leads to arterial dysfunction. This study will determine whether physiological shear-stress affects autophagosome formation and nitrous oxide (NO) generation in ECs.

DETAILED DESCRIPTION:
It is hypothesized that genetic autophagy suppression prevents shear-stress induced purinergic signaling to endothelial nitrous oxide synthase (eNOS) and this pathway will be evaluated in primary arterial ECs obtained from older adult (> 60 years) and adult (18-30 years) subjects before and following rhythmic handgrip exercise that elevates brachial artery shear-rate similarly in both groups. ECs will be used to quantify markers of EC autophagy, eNOS activation, and NO generation. The study will also determine whether exercise-training attenuates the aging-associated decline in EC autophagy, and whether intact autophagy is required for training-induced vascular improvements. To evaluate this potential, it will be determined whether one-limb rhythmic handgrip exercise training by older adult (> 60 y) human subjects is sufficient to elevate basal and shear-induced EC autophagy initiation, eNOS activation, and NO generation vs. the contralateral sedentary limb. Results from this work have tremendous potential to reveal a new therapeutic target and approach for restoring / maintaining vascular function in the aging population.

ELIGIBILITY:
Inclusion criteria:

* Candidates must be between 18 and 90 y of age
* Candidates must be free of overt disease as assessed by a) medical history; b) standard blood chemistries (chem. 7 panel), c) ECG at rest; d) limb vascular examination (ankle-brachial BP index > 0.9); e) resting BP < 140/90 mmHg; and f) skinfold % body fat assessment.
* Subjects will have a body mass index (BMI) between 19 and 30 and have plasma glucose concentrations < 7.0 mmol/L under fasting conditions and < 11.1 mmol/L at 120 minutes of an oral glucose tolerance test (OGTT)

Exclusion criteria

* Candidates <18 or >90 y of age
* Candidates demonstrating abnormal ECG, ankle-brachial BP index <0.9, resting BP > 140/90
* Candidates demonstrating a BMI <19 or > 30
* Candidates demonstrating plasma glucose concentrations > 7.0 mmol/L under fasting conditions and > 11.1 mmol/L at 120 minutes of an oral glucose tolerance test (OGTT)
* Candidates demonstrating dyslipidemia (plasma total cholesterol > 240 mg/dl with LDL-cholesterol > 160 mg/dl)
* Candidates reporting a history of myocardial infarction, unstable cardiac ischemia, recent cardiac catheterization, carotid artery disease, transient ischemic attack
* Women taking hormone replacement therapy (HRT) currently or in the preceding year will be excluded from the proposed studies due to the direct vascular effects of HRT.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Change in biomarker beclin-1 after Rhythmic Handgrip Exercise | 60 min
Change in biomarker Atg3 after Rhythmic Handgrip Exercise | 60 min
Change in biomarker Atg5 after Rhythmic Handgrip Exercise | 60 min
Change in biomarker Atg7 after Rhythmic Handgrip Exercise | 60 min
Change in biomarker Lamp1 after Rhythmic Handgrip Exercise | 60 min
Change in biomarker Lamp2 after Rhythmic Handgrip Exercise | 60 min
Change in biomarker p62 after Rhythmic Handgrip Exercise | 60 min
Change in biomarker beclin-1 after chronic exercise training | 8 weeks
Change in biomarker Atg3 after chronic exercise training | 8 weeks
Change in biomarker Atg5 after chronic exercise training | 8 weeks
Change in biomarker Atg7 after chronic exercise training | 8 weeks
Change in biomarker Lamp1 after chronic exercise training | 8 weeks
Change in biomarker Lamp2 after chronic exercise training | 8 weeks
Change in biomarker p62 after chronic exercise training | 8 weeks

SECONDARY OUTCOMES:
Change in radial arterial diameter after Rhythmic Handgrip Exercise | 60 min
Change in radial arterial flow rate after Rhythmic Handgrip Exercise | 60 min
Change in biomarker p-eNOSS1177 after Rhythmic Handgrip Exercise | 60 min
Change in radial arterial diameter after chronic exercise training | 8 weeks
Change in radial arterial flow rate after chronic exercise training | 8 weeks
Change in biomarker p-eNOSS1177 after chronic exercise training | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- VA Medical Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon written request, a limited, de-identified, anonymized dataset will be created pursuant to the Data use Agreement. This DUA will limit use of the dataset and prohibit the recipient from taking steps to identify individuals whose data is included in the dataset. This dataset will be provided through a password-protected, machine-readable database format. Whenever possible, the dataset will be delivered through physical transfer of a storage medium.